CLINICAL TRIAL: NCT03407846
Title: Total Laparoscopic Hystrectomy Versus Total Abdominal Hystrectomy: the Effect of Learning Curve a Randomized Controlled Trial
Brief Title: Total Laparoscopic Hystrectomy Versus Total Abdominal Hystrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed abd elfatah elsenity, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Total laparoscopic hystrectomy
Record Dates: First submitted 2017-09-20; First posted 2018-01-23 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Effect of Learning Curve on Operative Time in TLH and Comparing it to TAH

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total laparscopic hystrectomy (Active Comparator)
  Interventions: Procedure: Hystrectomy
- Total abdominal hystrectomy (Experimental)
  Interventions: Procedure: Hystrectomy

INTERVENTIONS:
Procedure: Hystrectomy — Total laparscopic hystrectomy versus total abdominal hystrectomy

SUMMARY:
100 patient will be recruited for hystrectomy for benign cause and TLH will be copared to TAH and effect of learning curve will be assessed by comparing operative time between early and lat patients in TLH group

ELIGIBILITY:
Inclusion Criteria:

- Age. More than 40 Uterine size less than 14 weeks No contraindications for laparscopic surgery Benign cause for hystrectomy

Exclusion Criteria:

* virgins Malignancy

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07-22 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-09-22 (Estimated)

PRIMARY OUTCOMES:
Operative time | 2 years
  Time in both type of hystrectomy will be compared and learning curve will be assesd among TLH group by comparing early cases to late

SECONDARY OUTCOMES:
Blood loss, coplications, postoperative pain | 2 years
  Hb measurment , and visual scale for pain

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Kept with researcher as cds for patients